CLINICAL TRIAL: NCT01834274
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Active-Controlled, 24-Week Study to Evaluate the Efficacy and Safety of Daily Oral TAK-875 50 mg Compared With Sitagliptin 100 mg When Used in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Comparison of Fasiglifam (TAK-875) With Sitagliptin When Used in Combination With Metformin in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_310; 2013-000542-19 (EudraCT Number); U1111-1139-0467 (Registry Identifier: WHO UTN); DOH-27-0913-4426 (Registry Identifier: SANCTR (South Africa)); NMRR-13-518-16346 (Registry Identifier: NMRR (Malaysia)); PHRR140127-000165 (Registry Identifier: PHRR (Philippines))
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fasiglifam 50 mg (Experimental): Fasiglifam (TAK-875) 50 mg tablets, orally, once daily, Sitagliptin placebo-matching tablets, orally, once daily, and metformin stable dose ≥1500 mg (or maximum-tolerated dose), tablets, orally, daily for up to 24 weeks.
  Interventions: Drug: Fasiglifam (TAK-875); Drug: Sitagliptin Placebo; Drug: Metformin
- Sitagliptin 100 mg (Active Comparator): Sitagliptin 100 mg, tablets, once daily, TAK-875 placebo-matching tablets, orally, once daily, and metformin stable dose ≥1500 mg (or maximum-tolerated dose), tablets, orally, daily for up to 24 weeks.
  Interventions: Drug: Fasiglifam (TAK-875) Placebo; Drug: Sitagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Fasiglifam (TAK-875) — Fasiglifam (TAK-875) tablets
  Arms: Fasiglifam 50 mg
Drug: Fasiglifam (TAK-875) Placebo — Fasiglifam (TAK-875) placebo-matching tablets
  Arms: Sitagliptin 100 mg
Drug: Sitagliptin — Sitagliptin tablets
  Arms: Sitagliptin 100 mg
Drug: Sitagliptin Placebo — Sitagliptin placebo-matching tablets
  Arms: Fasiglifam 50 mg
Drug: Metformin — Metformin tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy of fasiglifam (TAK-875) plus metformin compared with sitagliptin plus metformin on glycemic control over a 24-week Treatment Period.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-875. TAK-875 is being tested to treat people who have type 2 diabetes. This study will look at glycemic control in people who take TAK-875 in addition to metformin.

The study will enroll approximately 620 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-875 50 mg
* Sitagliptin 100 mg

All participants will be asked to take one tablet at the same time each day throughout the study. All participants will be asked to self-monitor their blood glucose levels and document any increases in blood glucose or symptoms of hypoglycemia in a diary.

This multi-center trial will be conducted in the United States, Latin America, Europe and Asia. The overall time to participate in this study is up to 42 weeks and participants will make up to 15 visits to the clinic.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is male or female and 18 years of age or older with a historical diagnosis of type 2 diabetes mellitus (T2DM).
4. Meets one of the following criteria:.

   1. Has an HbA1c ≥8% and <10.5%, and has been on a stable daily dose of ≥1500 mg (or documented maximum tolerated dose (MTD)) of metformin for at least 8 weeks prior to Screening. This participant will immediately enter the Placebo Run-in Period according to Study Schedule A, or;
   2. Has an HbA1c ≥8% and <10.5%, and has been on a stable daily dose of <1500 mg of metformin without documented MTD for at least 8 weeks prior to Screening. After completing the Screening Visit, these participants will have their metformin dose immediately increased to ≥1500 mg (or MTD) for an 8- to 12-week Titration/Stabilization Period according to Study Schedule B. Following stable administration of metformin ≥1500 mg (or MTD) for 8 weeks, the participant must qualify for entry into the Placebo Run-in Period by completing the Week -3 procedures and have an HbA1c ≥8% and <10.5%.
5. Has had no treatment with anti-diabetic agents other than metformin within 8 weeks prior to Screening (Exception: if a participant has received other anti-diabetic therapy for ≤7 days within the 8 weeks prior to Screening).
6. Has a body mass index (BMI) ≤45 kg/m^2 at Screening.
7. Participants regularly using other, non-excluded medications must be on a stable dose and regimen for at least 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator. Note: Participants who require initiation of a chronically administered medication(s) due to a disease or condition diagnosed at Screening must be rescreened after the new regimen has been stabilized.
8. A female participant of childbearing potential who is sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
9. Is able and willing to monitor glucose with a sponsor-provided home glucose monitor and consistently record his or her own blood glucose concentrations in diaries.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening or has received an investigational anti-diabetic drug within the 3 months prior to Screening.
2. Has been randomized into a previous TAK-875 study.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, or sibling) or may consent under duress.
4. Has donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. Has a hemoglobin ≤12 g/dL (≤120 g/L) for males and ≤10 g/dL (≤100 g/L) for females at Screening.
6. Has systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥95 mm Hg at Screening Visit. (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement and decision will be made on the second measurement.)
7. Has history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage I squamous cell carcinoma of the skin is allowed.
8. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2 x upper limit of normal (ULN) at Screening.
9. Has a total bilirubin level >ULN at Screening. Exception: if a participant has documented Gilbert's Syndrome the participant will be allowed with an elevated bilirubin level per the investigator's discretion.
10. Has serum creatinine ≥1.5mg/dL (≥133μmol/L) if male or ≥1.4 mg/dL (≥124 μmol/L) if female and/or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m^2 at Screening.
11. Has uncontrolled thyroid disease as determined by the investigator.
12. Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. Has a history of pancreatitis.
14. Has a history of gastric banding or gastric bypass surgery within one year prior to Screening.
15. Has a known history of infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
16. Had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction (MI), unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior to or at Screening.
17. Has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to any component of TAK-875, metformin, or sitagliptin.
18. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
19. Has received excluded medications prior to Screening or is expected to receive excluded medications.
20. If female, is pregnant (confirmed by laboratory testing, ie, serum/urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. Is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
22. Has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (104):
- United States (44):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - Garden Grove, California
  - Modesto, California
  - San Diego, California
  - Thousand Oaks, California
  - Lakewood, Colorado
  - Hallandale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - North Miami, Florida
  - North Miami Beach, Florida
  - Pembroke Pines, Florida
  - Sanford, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Evans, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Council Bluffs, Iowa
  - Augusta, Kansas
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Carlisle, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Fort Mill, South Carolina
  - Laurens, South Carolina
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Austin, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Victoria, Texas
  - Salt Lake City, Utah
- Argentina (3):
  - Coronel Suárez, Buenos Aires
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Rosario, Santa Fe Province
- Canada (8):
  - Calgary, Alberta
  - Red Deer, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Etobicoke, Ontario
  - London, Ontario
  - Toronto, Ontario
- Croatia (5):
  - Karlovac
  - Krapinske Toplice
  - Slavonski Brod
  - Virovitica
  - Zagreb
- Hungary (5):
  - Budapest
  - Gödöllő
  - Kistarcsa
  - Sátoraljaújhely
  - Szeged
- Malaysia (6):
  - Kelantan, Kelantan
  - Kuala Lumpur, Kuala Lumpur
  - Seri Manjung, Perak
  - Taiping, Perak
  - Taiping, Perak, Perak
  - Putrajaya, Selangor
- Peru (2):
  - Ica
  - Lima
- Philippines (6):
  - Cebu City
  - Iloilo City
  - Marikina City
  - Pasig
  - Quezon City
  - West Fairview, Quezon City
- Poland (7):
  - Gdansk
  - Lodz
  - Oświęcim
  - Rzeszów
  - Sobótka
  - Wroclaw
  - Zgierz
- Russia (4):
  - Barnaul
  - Kemerovo
  - Novosibirsk
  - Saint Petersburg
- South Africa (4):
  - Bloemfontein, Free State
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Thailand (5):
  - Bangkoknoi, Bangkok
  - Rajathevee, Bangkok
  - Muang, Changwat Khon Kaen
  - Klongluang, Changwat Pathum Thani
  - Hat Yai, Changwat Songkhla
- Ukraine (5):
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Vinnytsia

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 sites in the United States and 1 site in Canada from 18 May 2013 (first patient to sign informed consent) to 05 March 2014.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitis were enrolled equally in 1 of 2 treatment groups, once a day fasiglifam 50 mg or Sitagliptin 100 mg in combination with metformin.
Groups:
- Fasiglifam 50 mg: Fasiglifam 50 mg tablets, orally, once daily, sitagliptin placebo-matching tablets, orally, once daily, and metformin stable dose ≥1500 mg (or maximum-tolerated dose), tablets, orally, daily for up to 24 weeks.
- Sitagliptin 100 mg: Sitagliptin 100 mg, tablets, once daily, fasiglifam placebo-matching tablets, orally, once daily, and metformin stable dose ≥1500 mg (or maximum tolerated dose), tablets, orally, daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg
Started | 50 | 46
Completed | 3 | 5
Not Completed | 47 | 41
Not completed — Study Termination | 41 | 38
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (7.14) | 55.1 (9.07) | 56.4 (8.17)
Age, Customized [Number; unit: participants]
  < 65 years | 41 | 41 | 82
  ≥ 65 years | 9 | 5 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 26 | 26 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 1 | 3
  Black or African American | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 42 | 37 | 79
  Multiracial | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 34 | 31 | 65
  Non-Hispanic or Latino | 15 | 15 | 30
  Not Available | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 1
  United States | 49 | 46 | 95
Height [Mean (Standard Deviation); unit: cm] | 168.7 (11.45) | 169.9 (10.79) | 169.3 (11.10)
Weight [Mean (Standard Deviation); unit: kg] | 87.50 (18.769) | 96.09 (19.295) | 91.62 (19.408)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.77 (6.112) | 33.13 (4.787) | 31.90 (5.614)
Baseline BMI Category [Number; unit: participants]
  < 30 kg/m^2 | 31 | 11 | 42
  ≥ 30 kg/m^2 | 19 | 35 | 54
Baseline Glycosylated Hemoglobin (HbA)1c Category [Number; unit: participants]
  < 9% | 27 | 28 | 55
  ≥ 9 % | 23 | 18 | 41
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10.075 (6.530) | 8.877 (5.942) | 9.501 (6.252)
Smoking Classification [Number; unit: participants]
  Never smoked | 38 | 29 | 67
  Current smoker | 7 | 9 | 16
  Ex-smoker | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 or final visit relative to Baseline. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Week 24
Population: All randomized participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 4 | 3
Percent | -0.63 (0.340) [-1.1 to -0.3] | -0.43 (0.208) [-0.6 to -0.6]

2. Secondary Outcome: Percentage of Participants With HbA1c <7% at Week 24
Description: The percentage of participants with glycosylated hemoglobin less than 7% after 24 weeks of treatment.
Time Frame: Week 24
Population: As pre-defined in the SAP, no summary is provided for the secondary efficacy endpoint incidence of HbA1c <7% at Week 24 due to the limited enrollment and study duration at the time of study termination.
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: The change between FPG collected at week 24 or final visit relative to Baseline. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Week 24
Population: All randomized participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 4 | 3
mmol/L | -0.22 (1.971) | 1.54 (5.087)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blinded study drug.
Description: Safety population included all randomized participants who received at least one dose of study drug.
Arm/Group | Fasiglifam 50 mg | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/46
Other Adverse Events (participants affected / at risk) | 4/50 | 5/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasiglifam 50 mg (N=50) | Sitagliptin 100 mg (N=46)
Chest pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fasiglifam 50 mg (N=50) | Sitagliptin 100 mg (N=46)
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 3
Sinusitis (Infections and infestations) | 2 | 1
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.